CLINICAL TRIAL: NCT05620680
Title: Study of CD7 CAR-T Cells in Adult Refractory and Recurrent T-cell Lymphoma/Leukemia
Brief Title: CD7 CAR-T Cells in T-cell Lymphoma/Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-017
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: T Lymphoblastic Leukemia/Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): CD7 CAR-T treatment group
  Interventions: Biological: CD7 CAR-T cells

INTERVENTIONS:
Biological: CD7 CAR-T cells — patient was subjected to 0.5-2×10^6 cells/kg of CD7 CAR- T

SUMMARY:
T-cell lymphoma/leukemia is a group of highly lethal diseases with a high relapse rate and poor prognosis. CD7 was proved to be widely expressed in T-cell malignant, which makes it a promising therapeutic target.

In this study we aim to test the safety and efficacy of CD7 CAR-T cells in T-cell lymphoma/leukemia.

DETAILED DESCRIPTION:
T-cell lymphoma accounts for 10%~15% of non-Hodgkin lymphoma in China. According to the World Health Organization (WHO), T-cell lymphoma was divided into the following subtypes: T-cell, NK cell lymphoma/leukemia. There were two major categories: anterior T-cell tumors and posterior thymic T-cell lymphomas, which originate from lymph nodes, extranodal tissue, or skin; mature or peripheral T-cell lymphomas.

Generally speaking, the relapse accounts for 50-60% after first-line treatment, while the remission rate with second-line treatment was extremely low. Collectively, there was an urgent need for new treatment modalities to improve the clinical outcomes of these patients.

CD7 is a transmembrane glycoprotein that plays an important role in T-cell and T-cell/B-cell interactions during early lymphoid development. The expression of CD7 persist from stem to mature T cells. CD7 was proved to be widely expressed in T-cell malignant, which makes it a promising therapeutic target.

In this study we aim to testify the safy and efficacy of CD7 CAR-T cells in T-cell lymphoma/leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (≥ 18 years old, ≤ 75 years old), gender is not limited;
2. The subject voluntarily participates in the research and signs the "Informed Consent" by himself or his legal guardian;
3. According to the National Comprehensive Cancer Network (NCCN) T lymphocytic lymphoma (2020.V1)/acute lymphoblastic leukemia (2020. V1) practice guidelines, diagnosed with T-cell lymphoma;
4. Meet the diagnostic criteria for relapsed/refractory T-cell lymphoma, including any of the following:

1) Failure to obtain CR at the end of induction therapy; 2) Patients who have obtained CR have blasts in peripheral blood or bone marrow (proportion >5%), or extramedullary diseases; 5. Have not received antibody therapy within 2 weeks before cell therapy; 6. ECOG score of 0-2; 7. The subject has no contraindications to peripheral apheresis; 8. Expected survival time of more than 3 months.

Exclusion Criteria:

1. Those who have a history of allergy to any of the ingredients in cell products;
2. Laboratory tests for the following: including but not limited to, total serum bilirubin≧ 1.5mg/dl; Serum ALT or AST greater than 2.5 times the upper limit of normal; Blood creatinine≧ 2.0mg/dl; Platelet count≦ 10×109/L;
3. Patients with cardiac insufficiency who belong to class III or IV according to the New York Cardiology Association (NYHA) cardiac function grading standards; or echocardiography with left ventricular ejection fraction (LVEF) < 50%;
4. Abnormal lung function, blood oxygen saturation under indoor air < 92%;
5. Myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other serious clinical heart disease within 12 months before enrollment;
6. Grade 3 hypertension with poor control of blood pressure with medication;
7. Patients with other advanced tumors (those who are assessed as stable after treatment of other tumors can be enrolled);
8. Previous head trauma, impaired consciousness, epilepsy, more serious cerebral ischemia or cerebral hemorrhage disease;
9. Known central nervous system leukemia (CNS2 or CNS3), resistance to intrathecal chemotherapy injections and/or ongoing head and/or spinal radiation therapy; Previous CNS history but has been effectively controlled to allow enrollment;
10. Patients with autoimmune diseases, immunodeficiency or other patients requiring immunosuppressant therapy;
11. presence of uncontrolled, active infection;
12. Have previously used any CAR-T cell product or other genetically modified T cell therapy;
13. Live vaccination within 4 weeks prior to enrollment;
14. HIV, HBV, HCV and TPPA/RPR infections, and HBV carriers;
15. Subject has a history of alcoholism, drug addiction or mental illness;
16. The subject has participated in any other clinical research within 3 months before joining this clinical study;
17. Female subjects have any of the following conditions: a) are pregnant/lactating; or b) have plans to become pregnant during the trial; or c) are of childbearing potential and unable to use effective contraception;
18. There are other circumstances in which the investigator believes that the subject is not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
TEAEs | From date of initial treatment to the 30 days after treatment
  Adverse events during treatment

SECONDARY OUTCOMES:
overall response rate | baseline and 8 weeks, up to 1 year
  the proportion of complete and partial response patients

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China